CLINICAL TRIAL: NCT00891839
Title: An Open-Label Study of Bendamustine Hydrochloride in Combination With Rituximab in the Treatment of Patients With Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Bendamustine Hydrochloride in Combination With Rituximab in Patients With Relapsed Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18083/2039/NL/US-CA
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine+Rituximab (Experimental): Patients receive bendamustine at 90 mg/m^2 intravenously (iv) on days 1 and 2, and 375 mg/m^2 of rituximab by iv on day 1 of each 28-day cycle. Six 28-day cycles were planned and up to 8 cycles permitted for patients who do not have progressive disease and who have not achieved a complete response (CR).
  Interventions: Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine at 90 mg/m^2 intravenously (iv) on days 1 and 2 of each 28-day cycle. Dosage calculations for bendamustine are based on the patient's body surface area (BSA) at baseline, using actual weight for calculations. If there is a 10% change in a patient's weight during treatment, the most recent weight is used to recalculate the BSA. The new BSA is used in determining the doses to be administered in any subsequent cycles.
  Other Names: bendamustine HCl; TREANDA®; CEP-18083
Drug: Rituximab — Patients receive 375 mg/m^2 of rituximab, administered by iv infusion on day 1 of every 28-day cycle of treatment. Dosage calculations for rituximab are based on the patient's BSA at baseline, using actual weight for calculations. If there is a 10% change in a patient's weight during treatment, the most recent weight is used to recalculate the BSA. The new BSA is used in determining the doses to be administered in any subsequent cycles.
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the combination of bendamustine and rituximab in patients with relapsed/refractory mantle cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically confirmed diagnosis of typical or atypical mantle cell lymphoma, except for blastoid type.
* documented relapsed/refractory mantle cell lymphoma.
* CD20 positive B cells in the lymph node biopsy or other lymphoma pathology specimen.
* adequate hematologic function according to specific trial parameters.
* bidimensionally measurable disease with at least 1 lesion measuring 2.0 cm or more in a single dimension, or the patient is in the leukemic phase of the disease.
* patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* patient has an estimated life expectancy of at least 3 months.
* women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* men not surgically sterile or who are capable of producing offspring must practice abstinence or use a barrier method of birth control, and must agree to continue use of this method for the duration of study drug treatment and for 30 days after participation in the treatment period.

Exclusion Criteria:

* has received more than 3 previous standard chemotherapy regimens.
* has the blastoid subtype of mantle cell lymphoma.
* documented history of central nervous system (CNS) lymphomatous involvement.
* a history of previous high-dose chemotherapy with allogeneic stem cell transplantation (history of autologous stem cell transplantation is allowed).
* previous treatment with bendamustine.
* has an active malignancy other than MCL, or has had a malignancy other than MCL within the past 3 years, except for controlled prostate cancer without evidence of bone metastases, localized bladder cancer, cervical carcinoma in situ, breast cancer in situ, or non-melanoma skin cancer.
* has New York Heart Association (NYHA) Class III or IV heart failure, arrhythmias or unstable angina, electrocardiographic evidence of active ischemia or active conduction system abnormalities, or myocardial infarction within the last 6 months.
* has serum creatinine of more than 2.0 mg/dL or creatinine clearance of less than 30 mL/min based on the Cockcroft-Gault method or from a 24-hour urine collection.
* does not have adequate hepatic organ function as evidenced by specific trial parameters.
* has known human immunodeficiency virus (HIV) infection.
* has active hepatitis B infection. Hepatitis B surface antigen must be tested.
* a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* has received corticosteroids within 28 days of study entry unless chronically administered (prednisone ≤20 mg/day) for indications other than lymphoma or lymphoma-related complications.
* any serious uncontrolled, medical or psychological disorder that would impair the ability of the patient to participate in or complete this study.
* any condition which places the patient at unacceptable risk or confounds the ability of the investigators to interpret study data.
* patient has received other investigational agent(s) within 28 days of study entry.
* patient has received chemotherapy within the prior 28 days.
* patient has a known hypersensitivity to bendamustine, mannitol, or rituximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (13):
- United States (11):
  - Teva Investigational Site 11, Fountain Valley, California
  - Teva Investigational Site 2, Los Angeles, California
  - Teva Investigational Site 35, Orlando, Florida
  - Teva Investigational Site 30, Lafayette, Indiana
  - Teva Investigational Site 20, Bethesda, Maryland
  - Teva Investigational Site 4, Hackensack, New Jersey
  - Teva Investigational Site 3, Buffalo, New York
  - Teva Investigational Site 43, Gettysburg, Pennsylvania
  - Teva Investigational Site 33, Bryan, Texas
  - Teva Investigational Site 41, Grapevine, Texas
  - Teva Investigational Site 23, Lynchburg, Virginia
- Canada (2):
  - Teva Investigational Site 6, Ottawa
  - Teva Investigational Site 7, Toronto

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-five patients were screened and all were enrolled.
Groups:
- Bendamustine+Rituximab: Participants receive bendamustine at 90 mg/m^2 intravenously (iv) on days 1 and 2, and 375 mg/m^2 of rituximab by iv on day 1 of each 28-day cycle. Six 28-day cycles were planned and up to 8 cycles permitted for patients who do not have progressive disease and who have not achieved a complete response (CR).
Period: Overall Study
Arm/Group | Bendamustine+Rituximab
Started | 45
Completed | 38 (completed treatment)
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Disease progression | 3

BASELINE CHARACTERISTICS:
Population: Safety
Arm/Group | Bendamustine+Rituximab
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 39
  More than one race | 0
  Unknown or Not Reported | 2
Weight [Mean (Standard Deviation); unit: kg] | 80.3 (13.59)
Height [Mean (Standard Deviation); unit: cm] | 172.7 (9.87)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.9 (0.20)
Ann Arbor Staging System of Lymphoma [Number; unit: participants] — * Stage I indicates that the cancer is located in a single region.
  * Stage II indicates that the cancer is located in two separate regions, and that both affected areas are confined to one side of the diaphragm.
  * Stage III indicates that the cancer has spread to both sides of the diaphragm, including one organ or area near the lymph nodes or the spleen.
  * Stage IV indicates diffuse or disseminated involvement of one or more extralymphatic organs, including any involvement of the liver, bone marrow, or nodular involvement of the lungs
  participants
    Stage I | 0
    Stage II | 4
    Stage III | 4
    Stage IV | 37
B-Symptoms [Number; unit: participants] — The presence of B symptoms is a marker for more advanced disease with systemic, rather than merely local, involvement.
  B symptoms include:
  * Fever greater than 38 °C. Pel-Ebstein fever, the classic intermittent fever associated with Hodgkin disease, occurs at variable intervals of days to weeks and lasts for 1-2 weeks before resolving. However, fever associated with lymphoma can follow virtually any pattern.
  * Drenching sweats, especially at night.
  * Unintentional weight loss of >10% of normal body weight over a period of 6 months or less.
  participants
    Present | 9
    Absent | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Response + Partial Response) at the End of Cycles 3 and 6 Using the 2007 International Working Group Criteria
Description: The International Working Group (IWG) criteria (Cheson et al 2007) for a complete response is a complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. A partial response is at least a 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, no increase should be observed in the size of other nodes, liver or spleen, and no new sites of disease should be observed.
  95% CIs are calculated using binomial exact method.
Time Frame: Month 3 (end of cycle 3), Month 6 (end of cycle 6)
Population: Safety population consisting of all participants treated with at least 1 dose of bendamustine HCL.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine+Rituximab
Number analyzed (Participants) | 45
percentage of participants
  end of Cycle 3 | 71 [55.7 to 83.6]
  end of Cycle 6 | 82 [68.0 to 92.0]

2. Secondary Outcome: Kaplan-Meier Estimate for Duration of Response
Description: Duration of response is defined as the time between the date of the first response to date of progression or death. Response is determined on the basis of the 2007 IWG criteria. A complete response is a complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. A partial response is at least a 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, no increase should be observed in the size of other nodes, liver or spleen, and no new sites of disease should be observed.
Time Frame: Day 1 up to Month 43
Population: Safety population of participants who had a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine+Rituximab
Number analyzed (Participants) | 37
months | 18.9 [13.3 to 35.3]

3. Secondary Outcome: Kaplan-Meier Estimate for Progression-Free Survival
Description: Progression-free survival is defined as the time from first exposure to study medication to disease progression or relapse, or death due to any cause. Progression is defined using the 2007 International Working Group criteria, as any new lesion or increase by at least 50% of previously involved sites from nadir.
Time Frame: Day 1 up to Month 45
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine+Rituximab
Number analyzed (Participants) | 45
months | 17.2 [13.2 to 24.0]

4. Secondary Outcome: Kaplan-Meier Estimate for Overall Survival
Description: Overall survival is defined as the time from first exposure to study medication to death, or to last date from adverse events, concomitant medications, vital signs, lost to follow-up, or last known alive, for overall survival censoring date.
Time Frame: Day 1 up to Month 57
Population: Safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine+Rituximab
Number analyzed (Participants) | 45
months | 38.4 [23.4 to NA] — Upper range not estimable as not enough participants died

5. Secondary Outcome: Shifts in Baseline to Post-Treatment in Positron Emission Tomography (PET)
Description: Participants had a whole-body PET at baseline and at the end of cycle 6 or the end-of-treatment visit. Negative PET refers to PET results showing no abnormal lymph nodes; conversely, positive PET refers to PET results showing abnormal lymph nodes.
Time Frame: Baseline (Days -30 to 0), post treatment (up to Month 9, 30 days following completion of therapy)
Population: Safety population of participants with PET data
Measure: Number; unit: participants
Arm/Group | Bendamustine+Rituximab
Number analyzed (Participants) | 38
participants
  Baseline Negative - Study Negative | 0
  Baseline Positive - Study Negative | 0
  Baseline Negative - Study Positive | 23
  Baseline Positive - Study Positive | 15

6. Secondary Outcome: Shifts in Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The ECOG scale is:
  * Grade 0: Fully active, able to carry on all pre-disease activities without restriction;
  * Grade 1: Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  * Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours;
  * Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  * Grade 4: Completely disabled. Cannot carry on any self-care. Confined to bed or Chair.
  The shift table compares baseline ECOG scores to the ECOG scores as of the last treatment visit.
Time Frame: Day 0 (baseline) up to Month 8
Population: Safety population. One participant dropped out prior to obtaining a post-treatment ECOG evaluation.
Measure: Number; unit: participants
Arm/Group | Bendamustine+Rituximab
Number analyzed (Participants) | 44
participants
  Improved | 8
  Stayed the same | 32
  Deteriorated | 4

ADVERSE EVENTS:
Time Frame: Day 1 up to Month 8
Description: Participants are counted only once in each preferred term category, and only once in each system organ class category and high-level term.
Arm/Group | Bendamustine+Rituximab
Serious Adverse Events (participants affected / at risk) | 18/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine+Rituximab (N=45)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Toxoplasmosis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sedation (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine+Rituximab (N=45)
Anaemia (Blood and lymphatic system disorders) | 10 (14)
Leukopenia (Blood and lymphatic system disorders) | 9 (12)
Lymphopenia (Blood and lymphatic system disorders) | 6 (9)
Neutropenia (Blood and lymphatic system disorders) | 21 (29)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (21)
Tachycardia (Cardiac disorders) | 6 (6)
Vision blurred (Eye disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 17 (32)
Diarrhoea (Gastrointestinal disorders) | 16 (26)
Dry mouth (Gastrointestinal disorders) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 31 (61)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 16 (27)
Asthenia (General disorders) | 5 (7)
Chest pain (General disorders) | 3 (6)
Chills (General disorders) | 7 (15)
Fatigue (General disorders) | 25 (36)
Infusion related reaction (General disorders) | 4 (8)
Mucosal inflammation (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 7 (12)
Pyrexia (General disorders) | 13 (24)
Cytokine release syndrome (Immune system disorders) | 5 (11)
Pneumonia (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 4 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 3 (4)
Neutrophil count decreased (Investigations) | 3 (4)
Weight decreased (Investigations) | 14 (15)
Decreased appetite (Metabolism and nutrition disorders) | 19 (25)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 11 (18)
Dysgeusia (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 8 (13)
Anxiety (Psychiatric disorders) | 3 (5)
Confusional state (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (22)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 6 (14)
Flushing (Vascular disorders) | 4 (5)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.